CLINICAL TRIAL: NCT06587074
Title: Features of the Clinical Course and Prognosis in Patients With Idiopathic Pulmonary
Brief Title: Features of the Clinical Course and Prognosis in Patients With Idiopathic Pulmonary Hypertension When Using Modern Strategies of Specific Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Russian Cardiology Research and Production Center (Other)
Responsible Party: Principal Investigator, Tamila V. Martynyuk, MD, PhD, Professor, Head of pulmonary hypertension department, Russian Cardiology Research and Production Center
Other Study IDs: SHAM-3232
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1
- Group 2

SUMMARY:
This study will be performed based on a retrospective analysis of the cases of 150-170 patients with IPAH observed at the Research Institute of Clinical Cardiology over the past 10 years, for a comparative assessment of the survival of groups of patients with IPAH diagnosed in the period 2004-2013 and 2014-2023.

The demographic, clinical, functional, hemodynamic characteristics of patients, comorbidity, blood biomarker levels, received PAH-specific and symptomatic therapy will be assessed in order to determine the clinical characteristics of patients with IPAH.

The prospective part of study will include 50 patients with IPAH.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years;
* verified diagnosis of IPAH

Exclusion Criteria:

* age under 18 years;
* Other etiology op PAH,
* ischemic heart disease confirmed by MSCT of the coronary arteries or coronary angiography;
* diseases of the musculoskeletal system that prevent 6MWT
* severe liver dysfunction (more than 9 points on the Child-Pugh scale, class C)
* severe renal dysfunction (CC less than 15 ml/min), need for hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IPAH diagnosed patients in 2004-2023
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Mortality in 3 years after diagnosed IPAH | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tamila V Martyunuk, Yes, Principal Investigator — Russian National Cardiology Research Center
Locations (1):
- Russian National Cardilogy Reasearch Center, Moscow, Russia